CLINICAL TRIAL: NCT01293058
Title: Study of Routs of Naloxone Administration for Opioid Overdosed Patients
Brief Title: Randomized Trial of Intranasal Versus Intravenous Naloxone in Level of Consciousness in Suspected Opioid Overdose
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Dr. Alireza Yousefy, Associate Professor of Medical Education, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ASD-1213-16
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2007-03

CONDITIONS: Morphinan Opioid Overdose
Keywords: opioid; overdose; naloxone; intranasal
MeSH Terms: conditions — Drug Overdose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous (Other): The investigators administered intravenous naloxone for our opioid overdose patients
  Interventions: Drug: Intravenous
- Intranasal (Other): The investigators administered intranasal naloxone for treatment of our patients
  Interventions: Drug: Intranasal naloxone

INTERVENTIONS:
Drug: Intranasal naloxone — spray naloxone, 0.4 mg/ each 4 minutes till increasing patient level of consciousness
  Arms: Intranasal
Drug: Intravenous — Amp naloxone, 0.4 mg / each 4 minutes till increasing patient level of consciousness
  Arms: Intravenous

SUMMARY:
The purpose of this study is to determine which route of administration is better for treatment of opioid overdosed patients

DETAILED DESCRIPTION:
In intravenous drug abusers (IDUs), as a result of previous intravenous substance abuse, the predictable difficult cannulate exist and cause the delay administration of antidote therapy. Additionally, IDUs are also at increased risk of carrying blood borne infections that could be transmitted to healthcare workers through needle stick injuries. The investigators aimed to compare intranasal administration of naloxone with intravenous route.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the range of 15-50 years old

  * Who were suspicious to opioid overdoses based on history and having clinical appearance such as miotic pupils with loss of consciousness
  * Give response to naloxone with increasing the level of consciousness

Exclusion Criteria:

* Not giving response to naloxone and suspicious to have another reason for loss of consciousness

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2007-03; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
level of consciousness | 4 min after naloxone administration
  The investigators evaluated the level of consciousness with Glasgow coma sclae 4 minutes after naloxone administration

SECONDARY OUTCOMES:
blood pressure | at 4 min after naloxone administration
  The investigators evaluated blood pressure 4 minutes after naloxone administration

CONTACTS AND LOCATIONS:
Overall Officials: Nastaran Izadi, A.Professor, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Noor university hospital, Isfahan, Isfahan, Iran

REFERENCES:
- See also: Isfahan university of medical sciences — http://mui.ac.ir